CLINICAL TRIAL: NCT01481740
Title: A Double Blind Randomized Controlled Trial of Phenylephrine for the Prevention of Spinal Induced Hypotension in Obese Parturients
Brief Title: Preventing Hypotension in Parturients With an Elevated Body Mass Index (BMI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4999-01460
Record Dates: First submitted 2011-07-22; First posted 2011-11-30 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Hypotension
Keywords: spinal induced hypotension; nausea and vomiting; cesarean delivery
MeSH Terms: conditions — Hypotension; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenylephrine bolus (Experimental)
  Interventions: Drug: Phenylephrine bolus
- Phenylephrine infusion (Experimental)
  Interventions: Drug: phenylephrine infusion

INTERVENTIONS:
Drug: Phenylephrine bolus — 10 ml of 100mcg/ml phenylephrine and placebo infusion
  Arms: Phenylephrine bolus
Drug: phenylephrine infusion — 60ml infusion of 100mcg/ml phenylephrine and placebo bolus
  Arms: Phenylephrine infusion

SUMMARY:
Previous research regarding the use of phenylephrine has excluded obese subjects (BMI >35). This subgroup of patients represents a large portion of the obstetric patient population locally and nationally. It is unclear whether previous research should be extrapolated to the obese patient population. This study is being done to compare the incidence of hypotension, intraoperative nausea and vomiting, and neonatal acidosis between obese patients who receive a prophylactic phenylephrine infusion versus those who receive phenylephrine boluses for the treatment of established hypotension. This study will help us determine whether using a phenylephrine infusion or a phenylephrine bolus is the best way to prevent/treat spinal induced hypotension during cesarean deliveries in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* ASA Physical Status I-II
* Non-laboring women
* Single gestations ≥ 36 weeks
* Obese women (Body Mass Index 35 - 55 kg/m2)
* Non-emergent CD under spinal anesthesia

Exclusion Criteria:

* Height < 5'0"
* Antiemetic drug use in the 24 hours prior to CD
* Allergy to phenylephrine, or any other standardized medication
* Hypertensive disease of pregnancy (i.e. mild & severe preeclampsia)
* Chronic hypertension receiving antihypertensive treatment
* Severe Cardiac disease in pregnancy with marked functional limitations
* Patients on Monoamine Oxidase Inhibitors or Tricyclic Antidepressants
* Subject enrollment in another study involving a study medication within 30 days of CD
* Any other physical or psychiatric condition which may impair their ability to cooperate with study data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD FRCPC, Principal Investigator — IWK Health Centre
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] George RB, McKeen DM, Dominguez JE, Allen TK, Doyle PA, Habib AS. A randomized trial of phenylephrine infusion versus bolus dosing for nausea and vomiting during Cesarean delivery in obese women. Can J Anaesth. 2018 Mar;65(3):254-262. doi: 10.1007/s12630-017-1034-6. Epub 2017 Dec 5. PMID 29209926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Started | 90 | 88
Completed | 79 | 81
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion | Total
Number analyzed (Participants) | 79 | 81 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (6) | 31 (5) | 31 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 81 | 160
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 54 | 56 | 110
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nausea and Vomiting
Time Frame: intraoperative 2-3 hours
Measure: Number; unit: participants
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Number analyzed (Participants) | 79 | 81
participants | 59 | 37

2. Primary Outcome: Incidence of Nausea and Vomiting
Time Frame: 2 hrs postoperative
Measure: Number; unit: participants
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Number analyzed (Participants) | 79 | 81
participants | 29 | 26

3. Primary Outcome: Incidence of Nausea and Vomiting
Time Frame: 24hrs postoperative
Measure: Number; unit: participants
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Number analyzed (Participants) | 79 | 81
participants | 26 | 28

4. Secondary Outcome: Incidence of Hypotension
Time Frame: intraoperative - predelivery
Measure: Number; unit: participants
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Number analyzed (Participants) | 79 | 81
participants | 59 | 22

5. Secondary Outcome: Incidence of Hypotension
Time Frame: intraoperative - postdelivery
Measure: Number; unit: participants
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Number analyzed (Participants) | 79 | 81
participants | 34 | 6

6. Secondary Outcome: Neonatal Acidosis
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: pH value
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Number analyzed (Participants) | 79 | 81
pH value | 7.27 (0.06) | 7.27 (0.07)

ADVERSE EVENTS:
Arm/Group | Phenylephrine Bolus | Phenylephrine Infusion
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/81
Other Adverse Events (participants affected / at risk) | 0/79 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No